CLINICAL TRIAL: NCT02017197
Title: Therapeutic Equivalence Between Branded and Generic Warfarin Sodium Tablets in Adult Patients With Atrial Fibrillation in Brazil - Crossover Randomized Controlled Equivalence Trial
Brief Title: Therapeutic Equivalence Between Branded and Generic WARFArin Tablets in Brazil
Acronym: WARFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Carolina Gomes Freitas, Graduate student (PhD), Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RCT 01 GW; U1111-1155-4833 (Registry Identifier: Universal Trial Number (UTN))
Record Dates: First submitted 2013-12-11; First posted 2013-12-20 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Atrial Fibrillation
Keywords: Therapeutic Equivalency; Warfarin; Drugs, Generic; Anticoagulants; Anticoagulants [Pharmacological Action]; Coumarins
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence A (Other): Phase 1 (run-in): Marevan®
  Phase 2: Marevan®
  Phase 3: generic warfarin #1
  Phase 4: generic warfarin #2
  Interventions: Drug: Marevan®; Drug: generic warfarin #1; Drug: generic warfarin #2
- Sequence B (Other): Phase 1 (run-in): generic warfarin #1
  Phase 2: generic warfarin #1
  Phase 3: Marevan®
  Phase 4: generic warfarin #2
  Interventions: Drug: Marevan®; Drug: generic warfarin #1; Drug: generic warfarin #2
- Sequence C (Other): Phase 1 (run-in): generic warfarin #1
  Phase 2: generic warfarin #1
  Phase 3: generic warfarin #2
  Phase 4: Marevan®
  Interventions: Drug: Marevan®; Drug: generic warfarin #1; Drug: generic warfarin #2
- Sequence D (Other): Phase 1 (run-in): Marevan®
  Phase 2: Marevan®
  Phase 3: generic warfarin #2
  Phase 4: generic warfarin #1
  Interventions: Drug: Marevan®; Drug: generic warfarin #1; Drug: generic warfarin #2
- Sequence E (Other): Phase 1 (run-in): generic warfarin #2
  Phase 2: generic warfarin #2
  Phase 3: Marevan®
  Phase 4: generic warfarin #1
  Interventions: Drug: Marevan®; Drug: generic warfarin #1; Drug: generic warfarin #2
- Sequence F (Other): Phase 1 (run-in): generic warfarin #2
  Phase 2: generic warfarin #2
  Phase 3: generic warfarin #1
  Phase 4: Marevan®
  Interventions: Drug: Marevan®; Drug: generic warfarin #1; Drug: generic warfarin #2

INTERVENTIONS:
Drug: Marevan® — Branded warfarin sodium tablets (manufacturer União Química Farmacêutica Nacional S/A, Brazil) by mouth; dose adjusted according to INR and medical judgement.
  Other Names: warfarin
Drug: generic warfarin #1 — Generic warfarin sodium tablets, manufacturer (União Química Farmacêutica Nacional S/A, Brazil), by mouth; dose adjusted according to INR and medical judgement.
Drug: generic warfarin #2 — Generic warfarin sodium tablets, manufacturer (Laboratório Teuto Brasileiro S/A, Brazil), by mouth; dose adjusted according to INR and medical judgement.

SUMMARY:
The purpose of this study is to assess whether the switch from branded to generic warfarin or between different generic warfarin tablets may cause fluctuation in the results of coagulation tests (International Normalized Rate, acronym INR) in patients, thus predisposing them to unnecessary risks.

DETAILED DESCRIPTION:
[Changes to the protocol made until the stage of the statistical analysis plan, before data analysis and also before unblinding.]

1. Objective

   1.1 Main Objective

   We aim to determine, through mean INR difference between formulations, whether there is therapeutic equivalency between the branded warfarin sodium (Marevan®) and the generic formulations in atrial fibrillation patients in Brazil.

   1.2 Specific Objective

   In order to achieve the objective, we aim to assess with each warfarin formulation :
   * Delta INR [new primary outcome];
   * mean INR [mean prothrombin time will not be analyzed since it will convey the same information as the mean INR];
   * mean dosage needed for anticoagulation [new outcome];
   * clinical events (the frequency of thromboembolic events, bleedings, deaths and adverse events);
   * the time in therapeutic range;
   * and compliance with treatment.
2. Hypothesis

   Our hypothesis is that the delta INR of patients when using the generic tablets of warfarin sodium does not differ by more than 0.49 (two-sided) from the mean INR obtained when using the branded formulation, thereby demonstrating therapeutic equivalence. We will also assess this same outcome to assess therapeutic equivalence between the generic formulations to each other.
3. Type of Study

   This study is a crossover randomized controlled equivalence trial. It comprises four phases, each one one-month long, being the first one a run-in period. Patients will use a different warfarin sodium tablet formulation in each one of the phases 2, 3 and 4: either the branded Marevan® (União Química/Farmoquímica, Brasil), or two generic drugs, (manufactured by União Química Farmacêutica Nacional S/A or Laboratório Teuto Brasileiro S/A, Brasil) purchased from Brazilian drugstores (not directly from the manufacturer). Every patient will use each one of the three formulations in a previously determined sequence (A, B, C, D, E or F) to which he was assigned by randomization.

   Since patients included in the study will already be using warfarin and it is not ethically acceptable to interrupt this treatment, we planned a run-in period equivalent to seven warfarin half-lives, long enough to washout any previous warfarin treatment. Then, in this first phase, patients will start treatment with the same warfarin formulation that will be used in the second phase thus avoiding the carry-over effect. This period will also be used to select patients compliant with treatment, accepting those that during the run-in have at least one of the three (including the baseline) INR results within 2.0 and 3.0 and a difference of INR results at the 3th and 4th week ≤ ±0.8.
4. Methods

   An independent investigator (initials TFCP) will use a computer random number generator to allocate patients to one of the six sequences of treatment [update: we opted to apply randomization through numbered, opaque, sealed envelopes in order to facilitate allocation concealment]. The principal investigator (initials CGF) will separate, repack and dispense drugs for patients in opaque drug containers of identical appearance [update: the step of repacking the drugs in opaque containers was made by two investigators external to the study, BR and MFST, instead of the principal investigator]. This process will be based on the initials of the patient and the alphanumeric code, maintaining the allocation concealment since TFCP will be responsible for assigning to the repacked drugs the patient initials and the alphanumeric code correlated with the formulation of warfarin utilized. TFCP will also be accountable to conceal the allocation until the statistical analysis at the end of the study [update: BR and MFST created the coding and maintained its concealment]. Due to the features of the drug containers, physicians and the principal investigator (that assess patients and collect outcomes) will be blinded. Patients may not be blinded depending on the appearance of the manufactured tablets, but the main outcome will be a laboratory result (INR).
5. Sample Size

   Forty-eight patients (eight in each group) is the minimum necessary number of individuals to detect a clinically significant fluctuation of 0.49 in the mean INR, with a 90% power at a 5% level of significance, if one were present. This sample size was estimated considering the Pocock's statistical method for quantitative outcomes and an achieved mean INR and standard deviation with the branded warfarin of 2.45 and 0.29 respectively [update: later we considered a more conservative standard deviation of 0.34, which resulted in a sample size of 11 patients per group]. To compensate possible withdrawals or exclusions of patients we plan to recruit 60 patients.
6. Statistical Analysis

   For the INR, PT and TTR outcomes paired t-test will be used at a two-sided 5% level of significance. These analysis will be per protocol, i.e., data from patients that during the follow-up start treatment with substances or drugs that interact either in a moderate or major way or are contraindicated when used with warfarin (Annex I) will be excluded [update: multiple t-tests would not be adequate because nominal significance levels would not reflect the actual alfa, and thus we decided to apply multilevel mixed-effects linear regression. We have new definitions for per protocol analyses.].

   Binary outcomes (thromboembolic or bleeding events) will be analysed by Mcnemar test at a 5% level of significance using intention to treat i.e. considering missing data as adverse outcomes. In this case sensibility analysis will be conducted [update: we decided for just presenting the events recorded during the trial without any hypothesis testing due to cross-over design limitations and lower power for these outcomes]. Exploratory analysis for subgroup of patients are not intended.
7. Annex I (obtained from the online database Micromedex ® 2.0 in September 13, 2013)

   * abciximab
   * acarbose
   * acemetacin
   * acenocoumarol
   * acetaminophen
   * agrimony
   * alclofenac
   * alefacept
   * allopurinol
   * aloe
   * aminoglutethimide
   * amiodarone
   * amitriptyline
   * amobarbital sodium
   * amoxapine
   * amoxicillin
   * ampicillin trihydrate
   * amprenavir
   * angelica
   * anise
   * antithyroid agents
   * apazone
   * apixaban
   * aprepitant
   * aprobarbital
   * argatroban
   * armodafinil
   * arnica
   * asafetida
   * aspirin
   * astragalus
   * atazanavir
   * atenolol
   * atovaquone
   * avocado
   * azathioprine
   * azithromycin
   * bee pollen
   * benoxaprofen
   * benzbromarone
   * betamethasone
   * bicalutamide
   * bilberry
   * bismuth subsalicylate
   * bivalirudin
   * black cohosh extract
   * black currant
   * black haw
   * black tea
   * bladderwrack
   * boceprevir
   * bogbean
   * boldo
   * borage
   * bosentan
   * bromelain
   * bromfenac
   * buchu
   * bufexamac
   * butabarbital
   * butalbital
   * capecitabine
   * capsaicin
   * carbamazepine
   * carbenicillin disodium
   * carboplatin
   * carprofen
   * cassia
   * cat's claw
   * cefadroxil
   * cefamandole
   * cefazolin sodium
   * cefdinir
   * cefepime
   * cefixime
   * cefoperazone
   * cefotaxime
   * cefotetan
   * cefpodoxime
   * ceftazidime
   * ceftibuten
   * ceftizoxime
   * ceftriaxone
   * celecoxib
   * celery
   * cephalexin
   * cephalothin sodium
   * cephapirin
   * chamomile
   * chaparral
   * chitosan
   * chloral hydrate
   * chloramphenicol
   * chlordiazepoxide
   * chlorotrianisene
   * chlorpromazine hydrochloride
   * cholestyramine
   * chondroitin
   * cimetidine
   * cinchona
   * ciprofloxacin
   * cisapride monohydrate
   * cisplatin
   * citalopram
   * clarithromycin
   * clofibrate
   * clomipramine hydrochloride
   * clopidogrel
   * clove
   * clove oil
   * cloxacillin benzathine
   * coenzyme Q10
   * colesevelam
   * contraceptives, combination
   * cortisone
   * cranberry juice
   * curcumin
   * cyclophosphamide
   * cyclosporine, modified
   * dabigatran
   * dabrafenib
   * dalteparin
   * danaparoid
   * danazol
   * dandelion
   * dapsone
   * darunavir
   * deferasirox
   * delavirdine
   * demeclocycline
   * desipramine
   * desvenlafaxine
   * devil's claw
   * dexamethasone
   * dexlansoprazole
   * dexmethylphenidate
   * diazoxide
   * diclofenac
   * dicloxacillin
   * diethylstilbestrol
   * diflunisal
   * dipyridamole
   * dipyrone
   * disopyramide
   * disulfiram
   * dong quai
   * dothiepin
   * doxepin
   * doxorubicin
   * doxycycline calcium
   * dronedarone
   * droxicam
   * duloxetine
   * enoxacin
   * enoxaparin
   * enteral nutrition
   * enzalutamide
   * eptifibatide
   * erlotinib
   * erythromycin acistrate
   * escitalopram
   * esomeprazole
   * eterobarb
   * ethacrynic acid
   * ethanol
   * ethchlorvynol
   * ethotoin
   * etodolac
   * etoposide
   * etravirine
   * etretinate
   * evening primrose oil
   * exenatide
   * ezetimibe
   * felbamate
   * fenbufen
   * fenofibrate
   * fenofibric acid
   * fenoprofen
   * fenugreek
   * feverfew
   * fish oil
   * floctafenine
   * flosequinan
   * fluconazole
   * fludrocortisone acetate
   * flufenamic acid
   * fluorouracil
   * fluoxetine
   * fluoxymesterone
   * flurbiprofen
   * flutamide
   * fluvastatin
   * fluvoxamine
   * fosamprenavir
   * fosaprepitant
   * garlic
   * gatifloxacin
   * gefitinib
   * gemcitabine
   * gemfibrozil
   * gemifloxacin
   * ginger
   * ginkgo
   * ginseng, siberian
   * glimepiride
   * glipizide
   * glucagon
   * glucosamine
   * glutethimide
   * glyburide
   * goldenseal
   * green tea
   * griseofulvin
   * guggul
   * halothane
   * heparin calcium
   * heptabarbital
   * hexobarbital sodium
   * high protein food
   * horse chestnut
   * horseradish
   * hydrocortisone
   * ibritumomab
   * ibuprofen
   * ifosfamide
   * imatinib
   * imipramine hydrochloride
   * indomethacin
   * indoprofen
   * infliximab
   * influenza virus vaccine
   * ipriflavone
   * isoniazid
   * isoxicam
   * itraconazole
   * ivacaftor
   * ivermectin
   * kava
   * ketoconazole
   * ketoprofen
   * ketorolac tromethamine
   * lactulose
   * lansoprazole
   * leflunomide
   * lepirudin
   * levamisole
   * levofloxacin
   * licorice
   * lopinavir
   * lornoxicam
   * lovastatin
   * lycium
   * marijuana
   * meadowsweet
   * mechlorethamine
   * meclofenamate
   * mefenamic acid
   * melatonin
   * meloxicam
   * menthol
   * mephobarbital
   * mercaptopurine
   * mesalamine
   * mesna
   * methandrostenolone
   * methicillin
   * methotrexate
   * methyl salicylate
   * methylphenidate
   * methylprednisolone acetate
   * methyltestosterone
   * metronidazole
   * miconazole
   * mifepristone
   * milnacipran
   * minocycline hydrochloride
   * mistletoe
   * mitotane
   * moricizine hydrochloride
   * motherwort
   * moxalactam
   * moxifloxacin
   * nabumetone
   * nafcillin
   * nalidixic acid
   * nandrolone
   * naproxen
   * nelfinavir
   * neomycin
   * nettle extract
   * nevirapine
   * niacin
   * nilutamide
   * nimesulide
   * norfloxacin
   * nortriptyline hydrochloride
   * noscapine
   * ofloxacin
   * omega-3-acid ethyl esters
   * omeprazole
   * onion oil
   * orlistat
   * oseltamivir
   * oxacillin
   * oxandrolone
   * oxaprozin
   * oxymetholone
   * oxyphenbutazone
   * oxytetracycline
   * pantoprazole
   * papaya
   * paramethasone
   * paroxetine
   * parsley
   * passionflower
   * pau d'arco
   * penicillin G
   * penicillin V benzathine
   * pentosan polysulfate sodium
   * pentoxifylline
   * phenindione
   * phenobarbital
   * phenprocoumon
   * phenylbutazone
   * phenytoin
   * phytonadione
   * piperacillin
   * piracetam
   * pirazolac
   * piroxicam
   * pirprofen
   * policosanol
   * pomegranate
   * poplar
   * posaconazole
   * prasugrel
   * prednisolone
   * prednisone
   * prickly ash
   * primidone
   * procarbazine
   * proguanil
   * propafenone hydrochloride
   * propoxyphene
   * propranolol
   * propyphenazone
   * proquazone
   * protriptyline
   * pumpkin seed
   * quassia
   * quetiapine
   * quinestrol
   * quinidine
   * quinine
   * rabeprazole sodium
   * raloxifene
   * ranitidine
   * red clover
   * rifabutin
   * rifampin
   * rifapentine
   * rifaximin
   * rilonacept
   * ritonavir
   * rivaroxaban
   * rofecoxib
   * romidepsin
   * ropinirole
   * rosuvastatin
   * roxithromycin
   * salicylates
   * saquinavir
   * sarsaparilla
   * saw palmetto extract
   * secobarbital
   * senega
   * sertraline
   * simvastatin
   * sitaxsentan
   * skullcap
   * sorafenib
   * soybean
   * spironolactone
   * st john's wort
   * stanozolol
   * sucralfate
   * sulfamethoxazole
   * sulfasalazine
   * sulfinpyrazone
   * sulfisoxazole
   * sulindac
   * sulofenur
   * suprofen
   * sweet woodruff
   * tamarind
   * tamoxifen
   * tan shen
   * teduglutide
   * telaprevir
   * telithromycin
   * tenidap sodium
   * tenoxicam
   * terbinafine
   * teriflunomide
   * testosterone
   * tetracycline
   * thyroid hormones
   * tiaprofenic acid
   * tibolone
   * ticarcillin
   * ticlopidine
   * tigecycline
   * tinidazole
   * tinzaparin
   * tirofiban
   * tocilizumab
   * tolmetin
   * tolterodine tartrate
   * tonka
   * toremifene citrate
   * torsemide
   * tramadol
   * trastuzumab
   * treprostinil
   * triamcinolone acetonide
   * trimipramine
   * valdecoxib
   * valproic acid
   * vancomycin
   * vemurafenib
   * venlafaxine
   * vilazodone
   * vincristine
   * vindesine
   * vitamin A
   * vitamin E
   * vitamin K
   * voriconazole
   * vorinostat
   * wild lettuce
   * willow
   * wintergreen
   * yarrow
   * zafirlukast
   * zileuton
   * zomepirac sodium
   * zotepine

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of nonvalvular atrial fibrillation atrial flutter by electrocardiogram and echocardiography;
* CHA2DS2VASc score equal to or greater than 1;
* already in use of warfarin for at least 2 months;
* during the run-in, at least one of the three (including the baseline) INR results within 2.0 and 3.0 and a difference of INR results at the 3th and 4th week ≤ ±0.8
* signing of Informed Consent Form.

Exclusion Criteria:

* patients with serious contraindications to the use of anticoagulants (significant bleeding, known sensitivity to warfarin);
* women of childbearing age, pregnant or breastfeeding;
* patients with thrombocytopenia;
* patients with hepatic or renal impairment;
* patients with a history of bleeding episodes due to congenital deficiency of coagulation factors;
* patients enrolled in another trial;
* patients initiating treatment with drugs with major interactions or which are contraindicated when used concomitantly with warfarin, according to our list (Annex I).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Difference between Delta INR | At the fourth week of each period
  INR: International normalized ratio. INR will be assessed twice a month during the 16 weeks of study.
  Delta INR will be calculated by the difference, in absolute numbers (i.e. in module), between the two valid INR measurements due for each patient with each formulation at each period. Difference between the delta INRs will be the outcome. We will compare generic to branded warfarin (Marevan®) and the generic formulations to each other.

SECONDARY OUTCOMES:
Difference between mean INR | At the fourth week of each period
  INR: International normalized ratio. INR will be assessed twice a month during the 16 weeks of study.
  We will calculate the mean INR for each formulation of warfarin; difference between the mean INRs will be the outcome. We will compare generic to branded warfarin (Marevan®) and the generic formulations to each other.
Difference in warfarin dosage needed | At the fourth week of each period
  The warfarin dosage will be calculated as the sum of the dosage taken in the week before the study visit, as referred by the patient. We will calculate the mean dosage for each formulation of warfarin; difference between the mean dosage will be the outcome.
  We will compare generic to branded warfarin (Marevan®) and the generic formulations to each other.
Incidence of thromboembolic events | At the fourth week of each period
  Includes ischemic stroke (differential diagnosis with hemorrhagic stroke by tomography) and thromboembolism of viscera or extremities (diagnosed by acute symptoms and relevant diagnostic tests).
Incidence of bleeding events | At the fourth week of each period
  Classified as major or minor bleeding events.
  Major: intracranial hemorrhage, fatal bleeding, bleeding resulting in hemoglobin loss equal to or greater than 2.0 g / L, hemorrhage requiring transfusion, bleeding in sensitive areas such as the retina or pericardium.
  Minor: all other bleeding.
Time in therapeutic range (TTR) | At the fourth week of each period
  TTR calculated by Rosendaal Method also known as linear interpolation method. We will calculate the mean TTR for each formulation of warfarin; difference between the mean TTRs will be the outcome.
  We will compare generic to branded warfarin (Marevan®) and the generic formulations to each other.

OTHER OUTCOMES:
Compliance with treatment | At the fourth week of each period
  Performed by counting of returned pills

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Gomes Freitas, BPharm, Principal Investigator — Federal University of Sao Paulo (UNIFESP)
Locations (1):
- Hospital São Paulo/Hospital Universitário da UNIFESP (University Hospital of UNIFESP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Gomes Freitas C, Walsh M, Coutinho EL, Vincenzo de Paola AA, Atallah AN. Examining therapeutic equivalence between branded and generic warfarin in Brazil: The WARFA crossover randomized controlled trial. PLoS One. 2021 Apr 1;16(4):e0248567. doi: 10.1371/journal.pone.0248567. eCollection 2021. PMID 33793580
- [Derived] Freitas CG, Walsh M, Atallah AN. Design and rationale for the WARFA trial: a randomized controlled cross-over trial testing the therapeutic equivalence of branded and generic warfarin in atrial fibrillation patients in Brazil. BMC Cardiovasc Disord. 2017 Jun 7;17(1):148. doi: 10.1186/s12872-017-0584-4. PMID 28592234